CLINICAL TRIAL: NCT06221501
Title: Safety and Efficacy of Perioperative Efgartigimod Combined With Thymectomy for Thymoma and Myasthenia Gravis: A Prospective, Single-arm Study
Brief Title: Perioperative Efgartigimod for Thymoma and Myasthenia Gravis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-374R
Record Dates: First submitted 2023-12-27; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Efgartigimod Alfa — Efgartigimod will be administered intravenously on Day (D)1, D8, D15, and D22 at a dose of 10 mg/kg according to the patient's weight (maximum infusion dose of 1200 mg) over approximately 1 hour for a total of 4 doses. Thymectomy will be performed on Day 9.

SUMMARY:
It is evidenced that efgartigimod can rapidly and significantly improve the symptoms of myasthenia gravis. The global multicenter clinical trials hace confirmed that efgartigimod is safe and well tolerated. Few case reports showed that perioperative efgartigimod combined with thymectomy was safe and feasible. However, there was no sufficient data on safety and efficacy of this regimen in the treatment for patients with myasthenia gravis and thymomas. Therefore, this trial aims to evaluate the efficacy and safety of perioperative efgartigimod and thymectomy for patients with myasthenia gravis and thymomas.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged ≥ 18 years and ≤ 75 years with expected survival time > 12 months;
2. Patients with systemic Myasthenia gravis;
3. AChR Antibody positive;
4. MGFA Type II- IV;
5. Clinical diagnosis of Neoplasm of thymus by enhanced chest CT (clinical stage: Masaoka-Koga Stage I-IVa);
6. Patients with American Society of Anesthesiologists (ASA) classification of 1-2;
7. Subjects have no dysfunction of major organs; blood routine, lung, liver, kidney function and cardiac function are basically normal; laboratory test indicators must meet the following requirements: Blood: White cells > 4.0 x 109/L, absolute count of neutrophils (ANC) ≥ 2.0 x 109/L, Thrombocyte count > 100 x 109/L, Hemoglobin > 90 g/L; Lung function: FEV1 ≥ 1.2 L, FEV1% ≥ 50% and DLCO ≥ 50%. Note: FEV1: Forced vital capacity measured value (liter). FEV1%:% of Forced vital capacity observed/predicted. DLCO%: measured/predicted value% of diffusion capacity of the CO in one breath; Liver function: Serum bilirubin less than 1.5 times the maximum normal value; ALT and AST less than 1.5 times the maximum normal value; Renal function: blood creatinine (SCr) ≤ 120 µmol/L, creatinine clearance (CCr) ≥ 60 ml/min;
8. Understand the study and sign the informed consent form.

Exclusion Criteria:

1. Patients whose imaging investigation suggests that the tumor has already had hematogenous metastasis (clinical stage: Masaoka-Koga IVb);
2. Patients with ocular muscular myasthenia gravis (OMG);
3. Patients who have received median sternotomy ;
4. Documented history of congestive cardiac failure; poorly controlled drug therapy on Anginal pain; electrocardiogram (ECG) documented transmural myocardial infarction; poorly controlled hypertensive; clinically significant heart valve disorders; or high-risk uncontrolled arrhythmia;
5. Patients with a loss of more than 5 Kg within the past month; severe uncontrolled systemic intercurrent illness such as active Infection or poorly controlled Diabetes mellitus; patients with combined Hemorrhagic disorder and Haemorrhagic diathesis; patients with abnormal coagulation function, having haemorrhagic diathesis or receiving thrombolysis or anticoagulant therapy; and patients with grade II-IV myelosuppression.
6. Serum pregnancy test positive or lactating females, as well as males and females of childbearing potential who are unwilling to take adequate contraception measures during treatment;
7. History of organ transplant (including autologous bone marrow Transplant and peripheral Stem cell transplant);
8. Patients with peripheral nervous system disorders or significant history of Mental disorder and central nervous system disorders;
9. Concurrent participation in other clinical investigators.
10. Patients who cannot tolerate one-lung ventilation in the Surgery; patients with severe cardiac complications, cardiovascular compensatory dysfunction, cardiac pacemaker implantation;
11. Patients with acute Inflammation due to bacterial, viral or other pathogenic microorganism Infection; known Immunodeficiency virus (HIV), Hepatitis B virus (HBV) or Hepatitis C virus (HCV) active Infection or known HIV seropositivity;
12. Patients who previously underwent Thoracic operation for Tuberculous pleurisy, Mesothelioma, Pulmonary disorder, diaphragmatic disease, ipsilateral Atelectasis involving one lobe or more than one lobe;
13. Serum IgG level < 6 g/L;
14. Received biologic agents such as rituximab or eculizumab within 6 months; IV Immunoglobulins or Plasma exchange within 1 month;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of the activity of daily living (ADL) score at the fourth visit from the baseline visit (first visit) | Baseline and 3 weeks after the first visit.
  The value was calculated by the ADL score at the fourth visit minus the ADL score at the first visit (baseline).

SECONDARY OUTCOMES:
Change of the ADL score at the second visit from the baseline visit (first visit) | Baseline and 1 day before surgery (always at the 1 week after the first visit).
  The value was calculated by the ADL score at the second visit minus the ADL score at the first visit (baseline).
Change of quantitative myasthenia gravis (QMG) score at the second visit from the baseline visit (first visit) | Baseline and 1 day before surgery (always at the 1 week after the first visit).
  The value was calculated by the QMG score at the second visit minus the QMG score at the first visit (baseline).
Change of myasthenia gravis composite (MGC) score at the second visit from the baseline visit (first visit) | Baseline and 1 day before surgery (always at the 1 week after the first visit).
  The value was calculated by the MGC score at the second visit minus the MGC score at the first visit (baseline).
Change of QMG score at the fourth visit from the baseline visit (first visit) | Baseline and 3 weeks after the first visit.
  The value was calculated by the QMG score at the fourth visit minus the QMG score at the first visit (baseline).
Change of MGC score at the fourth visit from the baseline visit (first visit) | Baseline and 3 weeks after the first visit.
  The value was calculated by the MGC score at the fourth visit minus the MGC score at the first visit (baseline).
Change of lgG-AChR level at the fourth visit from the baseline visit (first visit) | Baseline and 3 weeks after the first visit.
  The value (percent) was calculated by the lgG-AChR level at the fourth visit minus the lgG-AChR level score at the first visit (baseline).
The rate of postoperative myasthenia crisis | From the day when trial begin to the day when the follow-up is ended. Up to 48 weeks.
Postoperative hospital stay | From the day when trial begin to the day when the follow-up is ended. Up to 48 weeks.

REFERENCES:
- [Derived] Wang S, Zhu M, Dong J, Zhang Y, Luo S, Jiang J, Cheng Z, Li Z, Yang W, Yu Y, Liu Z, Fan J, Xu X, Liu P, Zhang Z, Can F, Liang F, Jiang X, Tan L, Ding J. Perioperative Safety and Efficacy of Efgartigimod for Thymoma-Associated Myasthenia Gravis: A Prospective, Multicenter, Phase II Clinical Trial. J Thorac Oncol. 2025 Aug;20(8):1120-1130. doi: 10.1016/j.jtho.2025.04.014. Epub 2025 May 2. PMID 40320172